CLINICAL TRIAL: NCT05231213
Title: Effects of Neuromodulation and Cognitive Training for Suicide in Veterans (ENACTS)
Acronym: ENACTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4104-P
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Suicide; Impulsivity
Keywords: Suicide; Impulsive Behavior
MeSH Terms: conditions — Suicide; Impulsive Behavior

STUDY DESIGN:
Intervention Model Description: This study will be a double-blind, randomized, placebo (sham) controlled feasibility study. Thirty-eight Veteran inpatients in the Minneapolis VA Psychiatric unit will be recruited. Each participant will be randomly assigned to receive either active or sham tDCS, both paired with executive function cognitive training tasks. Training/tDCS sessions will occur twice a day for five days, for a total of 10 sessions. tDCS (2mA current), with anode over left prefrontal cortex and cathode over right prefrontal cortex, will be applied concurrently with cognitive training. Training/tDCS sessions last approx. 45 min, with tDCS applied during the first 20 min of training.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active tDCS (Experimental): Participants will receive 10 sessions of cognitive training concurrent with transcranial direct current stimulation (anode over left frontal cortex, cathode over right frontal cortex; 2 mAmps for 20 minutes).
  Interventions: Device: Active Transcranial Direct Current Stimulation (tDCS)
- Sham tDCS (Sham Comparator): Participants will receive 10 sessions of cognitive training concurrent with sham tDCS. For sham tDCS, electrodes are placed at the same locations as for active tDCS, but current is ramped up for the initial 30 secs, then immediately ramped back down. This method mimics the initial physical sensation of stimulation, but there is no active current for the remainder of the session.
  Interventions: Device: Sham Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Active Transcranial Direct Current Stimulation (tDCS) — Cognitive training concurrent with 2 mAmps of anodal stimulation applied to the left frontal cortex for 20 minutes.
  Arms: Active tDCS
Device: Sham Transcranial Direct Current Stimulation (tDCS) — Cognitive training concurrent with sham tDCS (30 secs ramp up/ramp down of current at beginning and end of session).
  Arms: Sham tDCS

SUMMARY:
Impaired executive function, such as impaired decision making and impulsivity, has been identified as an important contributor to the transition from suicidal ideation to suicide attempt. To address the epidemic of Veteran suicide in the United States, this study tests the feasibility, acceptability, and preliminary effectiveness of a five day transcranial direct current stimulation (tDCS) augmented executive functioning training intervention. This intervention is delivered to high suicide risk inpatients. The ultimate goal is to reduce future suicide events (ideation, attempts, deaths) and improve quality of life (e.g. social relationships, health resource utilization).

ELIGIBILITY:
Inclusion Criteria:

* currently admitted into the MVAHCS Inpatient Psychiatric Unit
* at a heightened risk for suicide (defined as a positive screen on the VA Comprehensive Suicide Risk Evaluation (CSRE) at intake and/or a suicide attempt within the previous 12 months)
* able to complete procedures and tasks

Exclusion Criteria:

* are unable to provide informed consent as determined by the Modified Dysken Tool
* have moderate/severe cognitive impairment as determined by the Mini-Mental State Examination (score 27)
* have contraindications for tDCS (history of seizures, metallic cranial plates/screws or implanted device, history of eczema on scalp)
* do not have a smartphone or device running Android or Apple iOS with which to download the mPRO EMA app
* have been involuntarily committed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Recruitment Feasibility | 2 years
  Recruitment feasibility will be demonstrated by successful recruitment of 15 participants per year into the study.
Intervention Acceptability | 2 months
  Acceptability of the intervention will be demonstrated by a retention rate of 80% at the 2 month follow-up assessment, and 70% of subjects tolerating the intervention (able to complete 2/3 of the twice-daily EMA surveys).

SECONDARY OUTCOMES:
Groton Maze Task | Change between baseline and 1 week follow-up; 1 and 2 months following intervention
  Differences in magnitude of change in performance on the Groton Maze Task between active and sham tDCS groups from baseline to follow-up sessions. Outcome score is time to complete task, with longer time indicating worse performance.
NIH Quality of Life questionnaire | Change between baseline and 1 week follow-up; 1 and 2 months following intervention
  Differences in magnitude of change in scores on the NIH Quality of Life (QOL) battery in the domains of cognitive, social, emotional, and behavioral abilities between active and sham tDCS groups from baseline to follow-up sessions. Responses are on a 0-5 Likert scale. Higher scores indicate better QOL.
UPPS-P Impulsive Behavior scale | Change between baseline and 1 week follow-up; 1 and 2 months following intervention
  The UPPS-P assesses impulsive behavior in five domains: Positive Urgency, Negative Urgency, (lack of) Premeditation, (lack of) Perseverance, and Sensation Seeking. The scale uses a 1 (agree strongly) to 4 (disagree strongly) response format. Higher scores indicate more impulsive behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Casey S Gilmore, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-11-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT05231213/ICF_000.pdf